CLINICAL TRIAL: NCT02708810
Title: RAD 1501: A Phase II Trial of Virtual Cone Trigeminal Neuralgia Radiosurgery
Brief Title: RAD 1501: A Trial of Virtual Cone Trigeminal Neuralgia Radiosurgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, John Fiveash, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-150608005
Record Dates: First submitted 2015-11-16; First posted 2016-03-15 (Estimated); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Trigeminal Neuralgia
Keywords: radiosurgery (RS); trigeminal neuralgia (TGN)
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Masks; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- 80 Gy Radiation & Unframed Virtual Cone (Other): 80 Gy Virtual Cone Radiosurgery unframed (face mask)
  Interventions: Device: Unframed Virtual Cone; Radiation: 80 Gy Radiation

INTERVENTIONS:
Device: Unframed Virtual Cone — A face mask (unframed) will be placed over the patient's face to keep their head from moving during the procedure. This will allow for very precise targeting. During the procedure, the study doctor will also confirm the exact location that needs to be treated using x-rays and optical imaging cameras. The face mask (unframed) will hold the patient's head to prevent it from moving and to focus the x-rays and aim them on the painful nerve in the patient's brain. For most patients, the actual time on the radiosurgery treatment machine is in the range of 30 to 60 minutes. The face mask (unframed) will be removed after the treatment.
  Other Names: Face Mask
Radiation: 80 Gy Radiation
  Other Names: Radiosurgery

SUMMARY:
To determine the feasibility of frameless Virtual Cone trigeminal neuralgia radiosurgery at a single institution prior to multi-institutional enrollment.

DETAILED DESCRIPTION:
To determine the feasibility of frameless Virtual Cone trigeminal neuralgia radiosurgery at a single institution prior to multi-institutional enrollment. To measure pain relief after Virtual Cone radiosurgery utilizing the Barrow Neurologic Institute Pain Intensity Score (BNI).

ELIGIBILITY:
Inclusion Criteria:

* Patients with trigeminal neuralgia pain that is not well controlled despite medical management (BNI 4 OR BNI 5)
* Patients must have an ECOG status of 0, 1, or 2
* Patients must be at least 18 years of age
* Life expectancy must be greater than 12 months
* MRI of brain within prior 12 months to confirm lack of other causes of facial pain
* All patients must be given written informed consent

Exclusion Criteria:

* Patients who have had prior brain radiosurgery or therapeutic radiation therapy to the pons
* Patients with atypical trigeminal neuralgia or headache pain syndromes
* Patients with pain associated with multiple sclerosis or base of skull tumor
* Patients with medical contra-indications to MR imaging (e.g. pacemaker)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Frameless Virtual Cone Trigeminal Neuralgia Radiosurgery as assessed by number of participants that completed treatment | 3 Month Follow-Up Visit
The mean of Barrow Neurologic Institute Pain Intensity Score (BNI) (pain relief score) between the two arms. | 1 Year
  Pain Relief Score designed to assess trigeminal neuralgia associated pain. It ranges from "I" being "no trigeminal pain, no medication" to "V" being "severe pain/no pain relief".

SECONDARY OUTCOMES:
Number of Participants with treatment-related adverse events | 1 Year
  Based on the assessments of the patient and the responses provided by the patient in questionnaires, we will assess acute and late neurologic toxicities. All adverse events/toxicities will be assessed with the utilization of CTCAE v.4.0.
Mean of Quality of Life Scores as measured by SF-36 Questionnaire | 1 Year
  Quality of Life (QOL) will be measured by SF-36. This questionnaire consists of 36 questions (items) measuring physical and mental health in relation to 8 health concepts: physical functioning, bodily pain, role of limitations due to physical health problems, role of limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perception. All items are scored so that a high score defines a more favorable health state. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are set at 0 and 100, respectively.
Patient Satisfaction Scores | 3 Month Follow-Up Visit
  3 months following the completion of radiosurgery, the patient will be asked the following two questions: 1) Would you have the radiosurgery procedure again? 2) Would you recommend it to friends and family?

CONTACTS AND LOCATIONS:
Overall Officials: John Fiveash, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Hazelrig-Salter Radiation Oncology Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No